CLINICAL TRIAL: NCT05364281
Title: The Changes of Endotracheal Tube Cuff Pressures While Positioning for Adenotonsillectomy or Tonsillectomy Surgery in Children: A Prospective Observational Study
Brief Title: The Changes of ETT Cuff Pressures After Head and Neck Positions Placed for Adenotonsillectomy and Tonsillectomy in Children
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Dilek Hundur, Attending Anesthesiologist, Istanbul University
Other Study IDs: 2019/155
Record Dates: First submitted 2022-05-04; First posted 2022-05-06 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2022-05

CONDITIONS: Endotracheal Tube Cuff Pressure; Adenotonsillectomy; Tonsillectomy; Position
Keywords: Pediatric Surgery; Endotracheal Tube Cuff Pressure; Adenotonsillectomy; Tonsillectomy; Position

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Patients younger than 18 years, who were scheduled for elective adenoidectomy or adenotonsillectomy operation.
  Interventions: Other: Intracuff pressure measurement

INTERVENTIONS:
Other: Intracuff pressure measurement — The intracuff pressures were measured and noted after each position (neck extension and placement of mouth gag), at every 5th minute while the operation and before the extubating.

SUMMARY:
The main purpose of this study was to assess the effect of each of position (neck extension by under-shoulder pillow and Crowe-Davis retractor use) during adenoidectomy and adenotonsillectomy on the intracuff pressure of ETTs in children.

DETAILED DESCRIPTION:
The cuff of the endotracheal tube seals the extraluminal airway to facilitate positive-pressure ventilation and reduce subglottic secretion aspiration. As increase or decrease of ETT intracuff pressures can lead to many morbidities. A total of 140 patients younger than 18 years, who were scheduled for elective adenoidectomy or adenotonsillectomy operation, were included in the study . A standardized general anesthetic was given and cuffed endotracheal tubes by the assistance of video laryngoscope were placed in all patients. The pilot balloon of each endotracheal tube was connected to the pressure transducer and standard invasive pressure monitoring was set to measure intracuff pressure values continuously. The first intracuff pressure value was adjusted to 18.4mmHg (25cm H2O) at supine and neutral neck position. The patients then were given appropriate position for the surgery. These positions were neck extension and placement of mouth gag These positions were neutral position, extension by under-shoulder pillow and placement of the mouth gag. The intracuff pressures were measured and noted after each position, at every 5th minute while the operation and before the extubating. If intracuff pressure deviated from the targeted value of 20-30cm H2O at any time, it was set to 25cm H2O again.

ELIGIBILITY:
Inclusion Criteria:

* Younger than 18 years
* American Society of Anesthesiologists (ASA) physical status I- II
* Elective tonsillectomy/ adenotonsillectomy under general anesthesia

Exclusion Criteria:

* Older than 18 years
* American Society of Anesthesiologists (ASA) physical status |>II
* Nasotracheal intubation
* Peroperative tracheotomy requirements
* Respiratory tract infection.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients younger than 18 years, who were scheduled for elective adenoidectomy or adenotonsillectomy operation, were included in the study .
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Intracuff Pressure | 0th minute (just after the positioning from neutral to surgical position)
  Endotracheal Tube Cuff Pressures in Adenotonsillectomy or Tonsillectomy Surgery Positions in Children

SECONDARY OUTCOMES:
Intracuff Pressure | From the beginning to the end of the operation before extubation
  Endotracheal Tube Cuff Pressure at every 5th minute while the operation and before the extubating

CONTACTS AND LOCATIONS:
Overall Officials: Emine Aysu Salviz, Assoc. Prof., Study Director — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Olsen GH, Krishna SG, Jatana KR, Elmaraghy CA, Ruda JM, Tobias JD. Changes in intracuff pressure of cuffed endotracheal tubes while positioning for adenotonsillectomy in children. Paediatr Anaesth. 2016 May;26(5):500-3. doi: 10.1111/pan.12873. Epub 2016 Mar 9. PMID 26956620